CLINICAL TRIAL: NCT00758758
Title: Performance of the Hedrocel(R) Cervical Fusion Device
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IC 003-99
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Symptomatic Cervical Disc Disease
Keywords: Anterior Cervical Discectomy and Fusion,; Degenerative Disc Disease,; Cervical Spine,; Herniated Disc
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Experimental Arm 1 (Experimental): Hedrocel 1 level - No plate
  Interventions: Device: Anterior Cervical Discectomy and Fusion
- Experimental Arm 2 (Experimental): Hedrocel 1 level with plate
  Interventions: Device: Anterior Cervical Discectomy and Fusion
- Experimental Arm 3 (Experimental): Hedrocel 2 levels with plate
  Interventions: Device: Anterior Cervical Discectomy and Fusion
- Control Arm 1 (Active Comparator): Autograft alone - Illiac crest
  Interventions: Device: Anterior Cervical Discectomy and Fusion
- Control Arm 2 (Active Comparator): Autograft 1 level with plate
  Interventions: Device: Anterior Cervical Discectomy and Fusion
- Control Arm 3 (Active Comparator): Allograft 1 level with plate
  Interventions: Device: Anterior Cervical Discectomy and Fusion
- Control Arm 4 (Active Comparator): Autograft 2 levels with plate
  Interventions: Device: Anterior Cervical Discectomy and Fusion
- Control Arm 5 (Active Comparator): Allograft 2 levels with plate
  Interventions: Device: Anterior Cervical Discectomy and Fusion

INTERVENTIONS:
Device: Anterior Cervical Discectomy and Fusion — Implantation of Hedrocel
  Arms: Experimental Arm 1; Experimental Arm 2; Experimental Arm 3
Device: Anterior Cervical Discectomy and Fusion — Implantation of Allograft
  Arms: Control Arm 3; Control Arm 5
Device: Anterior Cervical Discectomy and Fusion — Implantation of Autograft
  Arms: Control Arm 1; Control Arm 2; Control Arm 4

SUMMARY:
The objective of this clinical investigation is to compare patients treated with Anterior Cervical Discectomy and Fusion (ACDF) using the Hedrocel Cervical Fusion Device, with a concurrent, randomized, control group receiving autologous iliac crest bone graft or allograft and test the hypothesis that ACDF with Hedrocel is non-inferior to ACDF with allograft or autologous bone graft.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to compare patients treated with Anterior Cervical Discectomy and Fusion (ACDF) using the Hedrocel Cervical Fusion Device, with a concurrent, randomized, control group receiving autologous iliac crest bone graft. Success criteria include radiographic evidence of fusion, and improvement in pain, function and overall quality of life. If shown to be successful, the use of the Hedrocel Cervical Fusion Device would eliminate complications associated with harvesting autologous bone graft and provide an alternative for those who are unable to provide autologous bone graft from the iliac crest.

ELIGIBILITY:
Inclusion Criteria:

* The patient qualifies for ACDF based upon physical examination and medical history. The patient has single or two adjacent levels(s) symptomatic cervical disc disease (including disc herniation and/or spondylosis) from the C3-C4 disc to the C7-T1 disc with associated radiculopathy and/or myelopathy due to nerve root and/or spinal cord compression due to herniated nucleus pulposus or osteophyte formation on the posterior vertebral endplates. Patients who are candidates for surgery based on radicular symptoms must have at least one month of conservative treatment prior to inclusion in the study.
* The patient has no history of previous anterior cervical fusion surgery at the involved levels.
* The patient has no history of previous cervical fusion surgery at the adjacent levels.
* The patient is willing and able to provide written informed consent.
* The patient is likely to complete the required follow-up.

Exclusion Criteria:

* The patient is mentally compromised (e.g., under treatment for a psychiatric disorder or has senile dementia or Alzheimer's disease), or has evidence of alcohol or other substance abuse for the previous 12 months.
* The patient has a neuromuscular disorder that would engender unacceptable risk of instability, implant fixation failure, or complications in postoperative care.
* The patient has a diagnosed systemic disease that requires the chronic administration of nonsteroidal anti-inflammatory and steroidal drugs.
* The patient has osteopenia to a degree that would contraindicate spinal instrumentation (borderline osteoporosis).
* The patient has osteoporosis to a degree that would contraindicate spinal instrumentation.
* The patient is unable or unwilling to attend postoperative follow-up visits.
* The patient has received an investigational drug within the previous six months or an investigational device within the previous 12 months.
* The patient has a spinal condition other than Cervical DDD based upon physical examination and medical history.
* The patient has an infection site distant from the involved levels that may spread to the involved levels hematogenously.
* The patient has insufficient bone stock to fix the component.
* The patient has a known sensitivity to metallic implants.
* The patient is a prisoner.
* The patient has a Body Mass Index (BMI) greater than or equal to 40.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2001-12; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Cedars-Sinai Medical Center Institute for Spinal Disorders, Los Angeles, California
  - Orthopaedic Specialties, Clearwater, Florida
  - Southeastern Clinic Research, Orlando, Florida
  - Fort Wayne Orthopedics, Fort Wayne, Indiana
  - Spine Surgery PSC, Louisville, Kentucky
  - Four East Madison Orthopaedic Associates, PA, Baltimore, Maryland
  - Boston Spine Group, LLC, Boston, Massachusetts
  - Twin Cities Spine Center, Minneapolis, Minnesota
  - Orthocarolina, Charlotte, North Carolina
  - Howell Allen Clinic, Nashville, Tennessee
  - Vanderbilt Orthopedic Institute, Nashville, Tennessee
  - University of Virginia Health System - Department of Neurosurgery, Charlottesville, Virginia
  - Inova Fairfax Hospital, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between December 1999 and March 2007 from the investigators medical clinics.
Groups:
- Hedrocel 1 Level Without Plate: Hedrocel 1 level without plate
- Hedrocel 1 Level With Plate: Hedrocel 1 level with plate
- Hedrocel 2 Levels With Plate: Hedrocel 2 levels with plate
- Autograft Only - Illiac Crest: Autograft only - illiac crest
- Autograft 1 Level With Plate: Autograft 1 level plated
- Allograft 1 Level With Plate: Allograft 1 level plated
- Allograft 2 Levels With Plate: Allograft 2 levels with plate
- Autograft 2 Levels With Plate: Autograft 2 levels with plate
Period: Overall Study
Arm/Group | Hedrocel 1 Level Without Plate | Hedrocel 1 Level With Plate | Hedrocel 2 Levels With Plate | Autograft Only - Illiac Crest | Autograft 1 Level With Plate | Allograft 1 Level With Plate | Allograft 2 Levels With Plate | Autograft 2 Levels With Plate
Started | 14 | 74 | 53 | 6 | 3 | 50 | 31 | 0
Completed | 11 | 49 | 35 | 4 | 1 | 36 | 17 | 0
Not Completed | 3 | 25 | 18 | 2 | 2 | 14 | 14 | 0

BASELINE CHARACTERISTICS:
Groups:
- Autograft With Plate: Autograft with plate
- Allograft With Plate: Allograft with plate
- Total: Total of all reporting groups
Arm/Group | Hedrocel 1 Level Without Plate | Hedrocel 1 Level With Plate | Hedrocel 2 Levels With Plate | Autograft Only - Illiac Crest | Autograft With Plate | Allograft With Plate | Autograft 2 Levels With Plate | Allograft 2 Levels With Plate | Total
Number analyzed (Participants) | 14 | 74 | 53 | 6 | 3 | 50 | 0 | 31 | 231
Age Categorical [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Between 18 and 65 years | 14 | 74 | 53 | 6 | 3 | 50 |  | 31 | 231
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.14 (9.1) | 44.2 (8.6) | 49.0 (9.94) | 47.3 (5.0) | 49.0 (4.5) | 44.1 (6.8) |  | 49.29 (8.4) | 46.86 (7.5)
Gender [Number; unit: participants]
  Female | 3 | 43 | 28 | 2 | 0 | 25 |  | 20 | 121
  Male | 11 | 31 | 25 | 4 | 3 | 25 |  | 11 | 110
Region of Enrollment [Number; unit: participants]
  United States | 14 | 74 | 53 | 6 | 3 | 50 |  | 31 | 231

OUTCOME MEASURES:

1. Primary Outcome: Overall Clinical Success (NDI, Fusion, Additional Surgical Procedures)
Description: Success was defined as an improvement in patient functional capability using the Neck Disability Index (NDI) by at least 10% as compared to the pre-operative evaluation and Radiographic evidence of fusion (< 3mm translation; < 5° angular motion and absence of radiolucent lines around ≥ 50% of the device)and A comparison of the incidence of intraoperative and postoperative complications which resulted in additional surgical procedures of revision, removal or supplemental fixation at 12 months
Time Frame: 12 Months
Measure: Number; unit: participants
Groups:
- 1 Level Hedrocel Without Plate: 1 level Hedrocel with out plate
- One Level Hedrocel With Plate: Hedrocel with a plate
- Two Levels Plated Hedrocel: 2 Levels Plated Hedrocel
- Illiac Crest Autograft - no Plate: Iliac Crest Autograft
- Plated Autograft: Plated Autograft
- Plated Allograft: Plated Allograft
- 2 Levels Plated Autograft: 2 Levels with plated Autograft
- 2 Levels With Plated Allograft: 2 Levels with plated Allograft
Arm/Group | 1 Level Hedrocel Without Plate | One Level Hedrocel With Plate | Two Levels Plated Hedrocel | Illiac Crest Autograft - no Plate | Plated Autograft | Plated Allograft | 2 Levels Plated Autograft | 2 Levels With Plated Allograft
Number analyzed (Participants) | 11 | 49 | 35 | 4 | 1 | 36 | 0 | 17
participants | 5 | 33 | 28 | 2 | 1 | 22 |  | 15

2. Primary Outcome: Neck Disability Index (NDI)
Description: The Neck Disability Index (NDI) is an instrument used for testing self-rated disability in neck pain patients. The Neck Disability Index (NDI) consists of 10 questions, each with a score up to 5, for a total score of 50. The lower the score, the less self-rated disability.
  NDI scoring:
  * 0 - 4 = No disability
  * 5 - 14 = Mild disability
  * 15 - 24 = Moderate disability
  * 25 - 34 = Severe disability
  * 35 or over = Complete disability
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 1 Level Hedrocel Without Plate: 1 level Hedrocel without plate
- Hedrocel With Plate: Hedrocel with a plate
- 2 Levels Hedrocel With Plate: 2 Levels Plated Hedrocel
- Illiac Crest Autograft: Iliac Crest Autograft
- Autograft With Plate: Plated Autograft
- Allograft With Plate: Plated Allograft
- Autograft With 2 Plates: 2 Levels with plated Autograft
- Allograft With 2 Plates: 2 Levels with plated Allograft
Arm/Group | 1 Level Hedrocel Without Plate | Hedrocel With Plate | 2 Levels Hedrocel With Plate | Illiac Crest Autograft | Autograft With Plate | Allograft With Plate | Autograft With 2 Plates | Allograft With 2 Plates
Number analyzed (Participants) | 11 | 52 | 39 | 4 | 1 | 40 | 0 | 20
units on a scale | 14.82 (14.10) | 11.25 (10.30) | 8.77 (7.67) | 6.25 (8.02) | 1 (0) | 8.65 (8.56) |  | 10 (6.77)

ADVERSE EVENTS:
Arm/Group | Hedrocel 1 Level Without Plate | Hedrocel 1 Level With Plate | Hedrocel 2 Levels With Plate | Autograft Only - Illiac Crest | Autograft With Plate | Allograft With Plate | Autograft 2 Levels With Plate | Allograft 2 Levels With Plate
Serious Adverse Events (participants affected / at risk) | 2/14 | 2/74 | 1/53 | 0/6 | 0/3 | 0/50 | 0/0 | 1/31
Other Adverse Events (participants affected / at risk) | 2/14 | 9/74 | 15/53 | 0/6 | 0/3 | 5/50 | 0/0 | 2/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hedrocel 1 Level Without Plate (N=14) | Hedrocel 1 Level With Plate (N=74) | Hedrocel 2 Levels With Plate (N=53) | Autograft Only - Illiac Crest (N=6) | Autograft With Plate (N=3) | Allograft With Plate (N=50) | Autograft 2 Levels With Plate (N=0) | Allograft 2 Levels With Plate (N=31)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Fusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain- Neck and shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hedrocel 1 Level Without Plate (N=14) | Hedrocel 1 Level With Plate (N=74) | Hedrocel 2 Levels With Plate (N=53) | Autograft Only - Illiac Crest (N=6) | Autograft With Plate (N=3) | Allograft With Plate (N=50) | Autograft 2 Levels With Plate (N=0) | Allograft 2 Levels With Plate (N=31)
Device Loosening (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck and Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 7 (7) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint and muscle disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Surgical (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device Malfunction (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Numbness and Tingling (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Non-specific (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device Migration (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-Fusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less